CLINICAL TRIAL: NCT00129116
Title: A Phase II, Open (Partially Double-blind), Randomised, Controlled, Multicentre, Primary Vaccination Study to Evaluate the Immunogenicity, Reactogenicity and Safety of Three Different Formulations of GSK Biologicals' Combined Haemophilus Influenzae Type B-meningococcal Serogroups C and Y- Conjugate Vaccine and One Formulation of GSK Biologicals' Haemophilus Influenzae Type B-meningococcal Serogroup C Conjugate Vaccine Each Given Concomitantly With InfanrixTM Penta, Versus MeningitecTM, Given Concomitantly With InfanrixTM Hexa in Infants According to a 2-3-4 Month Schedule
Brief Title: 3 Formulations of Hib-MenCY-TT Vaccine & 1 Formulation of Hib-MenC-TT Vaccine Compared to Licensed Meningococcal Serogroup C Conjugate Vaccine, Each Administered at 2,3,4 Mths of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 792014/003; 100381 (Other: GSK)
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2016-10

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: Invasive bacterial disease caused by Hib; Neisseria meningitidis serogroups C & Y
MeSH Terms: conditions — Haemophilus Infections | interventions — Hib-MenCY-TT vaccine; DTPa-HBV-IPV combined vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- Menhibrix F1/Infanrix-penta Group (Experimental): Subjects received Menhibrix vaccine formulation 1 and Infanrix-penta vaccine. Vaccines were administered as a 3-dose primary vaccination course at 2, 3 and 4 months of age (at study Months 0, 1 and 2 of the primary phase). At 12-18 months of age (at study Month 0 of the booster phase), subjects received a booster dose of the two vaccines administered in the primary vaccination course. Menhibrix and Infanrix-penta vaccines were administered intramuscularly in the left and right anterolateral thigh, respectively.
  Interventions: Biological: Hib-MenCY-TT vaccine; Biological: Infanrix penta ®
- Menhibrix F2/Infanrix-penta Group (Experimental): Subjects received Menhibrix vaccine formulation 2 and Infanrix-penta vaccine. Vaccines were administered as a 3-dose primary vaccination course at 2, 3 and 4 months of age (at study Months 0, 1 and 2 of the primary phase). At 12-18 months of age (at study Month 0 of the booster phase), subjects received a booster dose of the two vaccines administered in the primary vaccination course. Menhibrix and Infanrix-penta vaccines were administered intramuscularly in the left and right anterolateral thigh, respectively.
  Interventions: Biological: Hib-MenCY-TT vaccine; Biological: Infanrix penta ®
- Menhibrix F3/Infanrix-penta Group (Experimental): Subjects received Menhibrix vaccine formulation 3 and Infanrix-penta vaccine. Vaccines were administered as a 3-dose primary vaccination course at 2, 3 and 4 months of age (at study Months 0, 1 and 2 of the primary phase). At 12-18 months of age (at study Month 0 of the booster phase), subjects received a booster dose of the two vaccines administered in the primary vaccination course. Menhibrix and Infanrix-penta vaccines were administered intramuscularly in the left and right anterolateral thigh, respectively.
  Interventions: Biological: Hib-MenCY-TT vaccine; Biological: Infanrix penta ®
- Menitorix/Infanrix-penta Group (Experimental): Subjects received Menitorix vaccine and Infanrix-penta vaccine. Vaccines were administered as a 3-dose primary vaccination course at 2, 3 and 4 months of age (at study Months 0, 1 and 2 of the primary phase). At 12-18 months of age (at study Month 0 of the booster phase), subjects received a booster dose of the two vaccines administered in the primary vaccination course. Menitorix and Infanrix-penta vaccines were administered intramuscularly in the left and right anterolateral thigh, respectively.
  Interventions: Biological: Hib-MenC-TT vaccine; Biological: Infanrix penta ®
- Menjugate/Infanrix-hexa Group (Active Comparator): Subjects received Menjugate vaccine and Infanrix-hexa vaccine. Vaccines were administered as a 3-dose primary vaccination course at 2, 3 and 4 months of age (at study Months 0, 1 and 2 of the primary phase). At 12-18 months of age (at study Month 0 of the booster phase), subjects received a booster dose of the two vaccines administered in the primary vaccination course. Menjugate and Infanrix-hexa vaccines were administered intramuscularly in the left and right anterolateral thigh, respectively.
  Interventions: Biological: Menjugate ®; Biological: Infanrix hexa ®

INTERVENTIONS:
Biological: Hib-MenCY-TT vaccine — Three doses during the primary vaccination and one booster dose administered intramuscularly (IM) in left thigh.
  Arms: Menhibrix F1/Infanrix-penta Group; Menhibrix F2/Infanrix-penta Group; Menhibrix F3/Infanrix-penta Group
Biological: Hib-MenC-TT vaccine — Three doses during the primary vaccination and one booster dose administered intramuscularly (IM) in left thigh.
  Arms: Menitorix/Infanrix-penta Group
Biological: Menjugate ® — Three doses during the primary vaccination and one booster dose administered intramuscularly (IM) in left thigh.
  Arms: Menjugate/Infanrix-hexa Group
Biological: Infanrix penta ® — Three doses during the primary vaccination and one booster dose administered intramuscularly (IM) in right thigh.
  Other Names: DTPa-HBV-IPV vaccine
  Arms: Menhibrix F1/Infanrix-penta Group; Menhibrix F2/Infanrix-penta Group; Menhibrix F3/Infanrix-penta Group; Menitorix/Infanrix-penta Group
Biological: Infanrix hexa ® — Three doses during the primary vaccination and one booster dose administered intramuscularly (IM) in right thigh.
  Other Names: DTPa-HBV-IPV/Hib vaccine
  Arms: Menjugate/Infanrix-hexa Group

SUMMARY:
This study evaluated the safety and immunogenicity of 3 formulations of Hib-MenCY-TT vaccine and 1 formulation of Hib-MenC-TT vaccine compared to a control group receiving licensed meningococcal serogroup C conjugate vaccine, each administered at 2, 3, and 4 months of age. Antibody persistence and immune responses to booster vaccinations were additionally assessed at 12 to 18 months of age.

DETAILED DESCRIPTION:
Primary & booster vaccination study to evaluate the immuno,reacto & safety of 3 diff. formulations of GSKBio'combined Haemophilus influenzae typeb-meningococcal serogroups C & Y-conjugate vaccine & one formulation of GSKBio' Haemophilus influenzae typeb-meningococcal serogroup C conjugate vaccine each given concomitantly With Infanrix penta (DTaP-IPV-HepB vaccine), vs Meningitec meningococcal SerogroupC conj.vaccine) given concomitantly With Infanrix hexa (DTaP-IPV-HepB-Hib vaccine) in infants according a 2-3-4 mth schedule

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants without major congenital illness, immunosuppression, or chronic disease born at 36 to 42 weeks of gestation, between 6 and 12 weeks of age at enrollment, and vaccinated against hepatitis B at birth.

Exclusion Criteria:

* Infants should not have received any investigational drug, vaccine, chronic immunosuppressants, or immunoglobulin or blood products.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 388 (Actual)
Dates: Start 2003-03-01; Primary Completion 2003-12-01 (Actual); Study Completion 2003-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- Belgium (7):
  - GSK Investigational Site, Asse
  - GSK Investigational Site, Drongen
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Maldegem
  - GSK Investigational Site, Merelbeke
  - GSK Investigational Site, Oudenaarde
  - GSK Investigational Site, Sint-Amandsberg
- Germany (14):
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Kaufering, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Niedernhausen, Hesse
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Kirchlengern, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bryant KA, Marshall GS. Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine for infants and toddlers. Expert Rev Vaccines. 2011 Jul;10(7):941-50. doi: 10.1586/erv.11.90. PMID 21806393
- [Background] Habermehl P, Leroux-Roels G, Sanger R, Machler G, Boutriau D. Combined Haemophilus influenzae type b and Neisseria meningitidis serogroup C (HibMenC) or serogroup C and Y-tetanus toxoid conjugate (and HibMenCY) vaccines are well-tolerated and immunogenic when administered according to the 2,3,4 months schedule with a fourth dose at 12-18 months of age. Hum Vaccin. 2010 Aug;6(8):640-51. doi: 10.4161/hv.6.8.12154. PMID 20697200
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 792014/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 792014/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 792014/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 792014/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 792014/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study is divided in two phases:
  * Primary phase: 3-dose primary vaccination at 2, 3 and 4 months of age = study Months 0, 1, 2. Data were collected up to 1 month after the 3rd dose (study Month 3)
  * Booster phase: booster dose at 12-18 months of age = study Month 0. Data were collected up to 1 month after the booster dose (study Month 1)
Period: Primary Phase
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Started | 78 | 77 | 78 | 78 | 77
Completed | 76 | 73 | 77 | 77 | 76
Not Completed | 2 | 4 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Period: Booster Phase
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Started | 47 | 42 | 44 | 44 | 44
Completed | 45 | 42 | 44 | 44 | 43
Not Completed | 2 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group | Total
Number analyzed (Participants) | 78 | 77 | 78 | 78 | 77 | 388
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.5 (1.69) | 8.8 (1.72) | 8.7 (1.55) | 8.3 (1.63) | 9.0 (1.65) | 8.7 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 37 | 44 | 33 | 40 | 185
  Male | 47 | 40 | 34 | 45 | 37 | 203

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Equal to or Above 1 Microgram Per Millilitre (µg/mL).
Description: Anti-PRP antibody concentration cut-off value assessed was equal to or above (≥) 1 microgram per millilitre (µg/mL)
Time Frame: One month after dose 3 (at study Month 3 - primary phase)
Population: The According-To-Protocol cohort for immunogenicity included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component, for at least one blood sample.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 67 | 67 | 70 | 74 | 71
Subjects | 66 | 66 | 69 | 73 | 57

2. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titre Equal to or Above 1:8
Description: rSBA-MenC antibody titre cut-off value assessed was ≥1:8
Time Frame: One month after dose 3 (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 70 | 67 | 71 | 74 | 71
Subjects | 70 | 67 | 71 | 74 | 71

3. Primary Outcome: Number of Subjects With Meningococcal Serogroup Y Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenY) Titre Equal to or Above 1:8
Description: rSBA-MenY antibody titre cut-off value assessed was ≥1:8
Time Frame: One month after dose 3 (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 66 | 71 | 74 | 71
Subjects | 67 | 64 | 70 | 16 | 14

4. Primary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Equal to or Above 1 Microgram Per Millilitre (µg/mL).
Description: Anti-PRP antibody concentration cut-off value assessed was equal to or above (≥) 1 microgram per millilitre (µg/mL)
Time Frame: One month after the booster vaccination (at study Month 1 - booster phase)
Population: The Booster According-To-Protocol cohort for immunogenicity included all vaccinated subjects who complied with the procedures defined in the protocol and for whom immunogenicity data were available.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 39 | 39 | 39 | 40 | 39
Subjects | 39 | 39 | 39 | 40 | 39

5. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titre Equal to or Above 1:8
Description: rSBA-MenC antibody titre cut-off value assessed was ≥1:8
Time Frame: One month after the booster vaccination (at study Month 1 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 40 | 39 | 42 | 41 | 39
Subjects | 40 | 39 | 42 | 41 | 39

6. Primary Outcome: Number of Subjects With Meningococcal Serogroup Y Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenY) Titre Equal to or Above 1:8
Description: rSBA-MenY antibody titre cut-off value assessed was ≥1:8
Time Frame: One month after the booster vaccination (at study Month 1 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 40 | 39 | 42 | 40 | 39
Subjects | 40 | 39 | 42 | 13 | 14

7. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titre Equal to or Above 1:8
Description: rSBA-MenC antibody titre cut-off value assessed was ≥1:8
Time Frame: Before the administration of the first dose (at pre-vaccination = study Month 0 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 64 | 70 | 73 | 71
Subjects | 4 | 6 | 4 | 6 | 3

8. Secondary Outcome: Number of Subjects With Meningococcal Serogroup Y Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenY) Titre Equal to or Above 1:8
Description: rSBA-MenY antibody titre cut-off value assessed was ≥1:8
Time Frame: Before the administration of the first dose (at pre-vaccination = study Month 0 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 70 | 63 | 71 | 73 | 71
Subjects | 11 | 10 | 16 | 10 | 17

9. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Equal to or Above 1 Microgram Per Millilitre (µg/mL).
Description: Anti-PRP antibody concentration cut-off value assessed was equal to or above (≥) 1 microgram per millilitre (µg/mL)
Time Frame: Before the administration of the first dose (at pre-vaccination = study Month 0 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 63 | 71 | 73 | 71
Subjects | 13 | 8 | 8 | 9 | 3

10. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Equal to or Above 1 Microgram Per Millilitre (µg/mL).
Description: Anti-PRP antibody concentration cut-off value assessed was equal to or above (≥) 1 microgram per millilitre (µg/mL)
Time Frame: Prior to the booster vaccination (at study Month 0 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 41 | 39 | 42 | 42 | 36
Subjects | 26 | 28 | 27 | 32 | 11

11. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titre Equal to or Above 1:8
Description: rSBA-MenC antibody titre cut-off value assessed was ≥1:8
Time Frame: Prior to the booster vaccination (at study Month 0 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 42 | 39 | 41 | 41 | 38
Subjects | 38 | 38 | 38 | 39 | 36

12. Secondary Outcome: Number of Subjects With Meningococcal Serogroup Y Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenY) Titre Equal to or Above 1:8
Description: rSBA-MenY antibody titre cut-off value assessed was ≥1:8
Time Frame: Prior to the booster vaccination (at study Month 0 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 41 | 39 | 42 | 42 | 37
Subjects | 35 | 31 | 36 | 11 | 15

13. Secondary Outcome: rSBA-MenC Antibody Titres
Description: Titres are expressed as geometric mean titres (GMTs)
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 70 | 67 | 71 | 74 | 71
Titers
  rSBA-MenC [Month 0] (N=69,64,70,73,71) | 4.7 [3.9 to 5.7] | 4.8 [4.1 to 5.6] | 4.6 [4.0 to 5.4] | 4.7 [4.0 to 5.7] | 4.5 [3.9 to 5.2]
  rSBA-MenC [Month 3] (N=70,67,71,74,71) | 1005.8 [773.5 to 1308.0] | 1029.8 [799.7 to 1326.0] | 906.9 [691.3 to 1189.8] | 871.0 [677.3 to 1120.0] | 3557.6 [2978.8 to 4248.8]

14. Secondary Outcome: rSBA-MenY Antibody Titres
Description: Titres are expressed as geometric mean titres (GMTs)
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 70 | 66 | 71 | 74 | 71
Titers
  rSBA-MenY [Month 0] (N=70,63,71,73,71) | 5.9 [4.7 to 7.5] | 5.9 [4.6 to 7.6] | 7.4 [5.6 to 9.9] | 5.9 [4.6 to 7.4] | 7.7 [5.7 to 10.3]
  rSBA-MenY [Month 3] (N=69,66,71,74,71) | 470.7 [351.1 to 631.2] | 437.1 [322.0 to 593.4] | 635.3 [501.5 to 804.8] | 9.3 [6.3 to 13.7] | 7.5 [5.4 to 10.4]

15. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Equal to or Above 0.15 Microgram Per Millilitre (µg/mL).
Description: Anti-PRP antibody concentration cut-off value assessed was equal to or above (≥) 0.15 microgram per millilitre (µg/mL)
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 67 | 71 | 74 | 71
Subjects
  Anti-PRP >= 0.15 µg/mL [Mth 0] (N=69,63,71,73,71) | 51 | 42 | 50 | 50 | 50
  Anti-PRP >= 0.15 µg/mL [Mth 3] (N=67,67,70,74,71) | 67 | 67 | 70 | 74 | 71

16. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in µg/mL.
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 67 | 71 | 74 | 71
µg/mL
  Anti-PRP [Month 0] (N=69,63,71,73,71) | 0.289 [0.217 to 0.385] | 0.243 [0.185 to 0.318] | 0.255 [0.197 to 0.331] | 0.243 [0.184 to 0.319] | 0.217 [0.177 to 0.267]
  Anti-PRP [Month 3] (N=67,67,70,74,71) | 9.014 [7.248 to 11.209] | 9.485 [7.721 to 11.651] | 8.075 [6.532 to 9.982] | 10.435 [8.487 to 12.830] | 2.595 [1.965 to 3.428]

17. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentration Equal to or Above 0.30 Microgram Per Millilitre (µg/mL)
Description: Anti-PSC antibody concentration cut-off value assessed was ≥0.30 µg/mL
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 66 | 71 | 74 | 71
Subjects
  Anti-PSC [Month 0] (N=69,63,71,74,71) | 7 | 12 | 7 | 7 | 10
  Anti-PSC [Month 3] (N=69,66,70,74,71) | 69 | 66 | 70 | 74 | 71

18. Secondary Outcome: Number of Subjects With Anti-polysaccharide Y (Anti-PSY) Antibody Concentration Equal to or Above 0.30 Microgram Per Millilitre (µg/mL)
Description: Anti-PSY antibody concentration cut-off value assessed was ≥0.30 µg/mL
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 66 | 71 | 74 | 71
Subjects
  Anti-PSY [Month 0] (N=69,64,71,73,71) | 7 | 6 | 12 | 15 | 12
  Anti-PSY [Month 3] (N=69,66,70,74,71) | 69 | 66 | 70 | 6 | 4

19. Secondary Outcome: Anti-PSC Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in µg/mL.
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 66 | 71 | 74 | 71
µg/mL
  Anti-PSC [Month 0] (N=69,63,71,74,71) | 0.18 [0.16 to 0.20] | 0.20 [0.17 to 0.24] | 0.18 [0.16 to 0.21] | 0.18 [0.15 to 0.22] | 0.18 [0.16 to 0.21]
  Anti-PSC [Month 3] (N=69,66,70,74,71) | 21.70 [18.36 to 25.65] | 27.26 [23.26 to 31.95] | 19.02 [16.49 to 21.93] | 21.08 [18.24 to 24.35] | 38.49 [33.64 to 44.05]

20. Secondary Outcome: Anti-PSY Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in µg/mL.
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 66 | 71 | 74 | 71
µg/mL
  Anti-PSY [Month 0] (N=69,64,71,73,71) | 0.19 [0.16 to 0.23] | 0.18 [0.15 to 0.20] | 0.20 [0.17 to 0.25] | 0.22 [0.18 to 0.27] | 0.20 [0.17 to 0.23]
  Anti-PSY [Month 3] (N=69,66,70,74,71) | 26.86 [22.86 to 31.56] | 37.02 [31.84 to 43.04] | 23.57 [19.94 to 27.86] | 0.19 [0.15 to 0.25] | 0.17 [0.15 to 0.19]

21. Secondary Outcome: Anti-tetanus Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in International Units per millilitre (IU/mL).
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 67 | 71 | 74 | 71
IU/mL
  Anti-tetanus [Month 0] (N=69,63,71,73,71) | 0.433 [0.320 to 0.586] | 0.485 [0.373 to 0.630] | 0.523 [0.388 to 0.705] | 0.436 [0.323 to 0.589] | 0.379 [0.285 to 0.503]
  Anti-tetanus [Month 3] (N=68,67,70,74,71) | 3.057 [2.629 to 3.554] | 3.254 [2.879 to 3.677] | 2.972 [2.591 to 3.409] | 3.151 [2.726 to 3.641] | 1.656 [1.394 to 1.967]

22. Secondary Outcome: Anti-filamentous Haemagglutinin (Anti-FHA), Anti-pertactin (Anti-PRN), Anti-pertussis Toxoid (Anti-PT) Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in Enzyme-Linked Immunosorbent Assay (ELISA) Units per millilitre.
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 67 | 71 | 74 | 71
EL.U/mL
  Anti-PT [Month 0] (N=67,62,68,70,69) | 3.4 [2.9 to 4.0] | 3.1 [2.7 to 3.5] | 3.7 [3.0 to 4.6] | 3.3 [2.8 to 4.0] | 3.1 [2.7 to 3.5]
  Anti-PT [Month 3] (N=67,63,69,74,69) | 53.9 [46.3 to 62.7] | 52.9 [45.3 to 61.8] | 50.8 [44.1 to 58.5] | 55.4 [48.1 to 63.7] | 41.3 [35.1 to 48.5]
  Anti-FHA [Month 0] (N=69,63,69,72,70) | 6.5 [5.2 to 8.1] | 6.0 [4.8 to 7.5] | 7.3 [5.7 to 9.3] | 9.9 [7.8 to 12.6] | 7.0 [5.6 to 8.7]
  Anti-FHA [Month 3] (N=67,63,69,74,71) | 83.7 [72.9 to 96.0] | 91.5 [78.7 to 106.3] | 89.3 [78.4 to 101.6] | 92.4 [79.8 to 106.9] | 74.0 [64.9 to 84.5]
  Anti-PRN [Month 0] (N=68,62,71,72,70) | 6.3 [4.9 to 8.2] | 4.5 [3.6 to 5.7] | 5.5 [4.5 to 6.8] | 6.4 [4.9 to 8.3] | 6.5 [5.0 to 8.4]
  Anti-PRN [Month 3] (N=68,67,70,74,71) | 94.2 [77.6 to 114.5] | 97.1 [79.8 to 118.2] | 96.2 [80.2 to 115.5] | 99.1 [79.0 to 124.3] | 80.2 [66.1 to 97.2]

23. Secondary Outcome: Number of Seroprotected Subjects for Anti-tetanus Antibodies
Description: Seroprotection status is defined as anti-tetanus toxoid antibody concentration ≥ 0.1 International Units per millilitre (IU/mL)
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 67 | 71 | 74 | 71
Subjects
  Anti-tetanus [Month 0] (N=69,63,71,73,71) | 58 | 57 | 60 | 63 | 61
  Anti-tetanus [Month 3] (N=68,67,70,74,71) | 68 | 67 | 70 | 74 | 71

24. Secondary Outcome: Number of Subjects With Anti-FHA, Anti-PRN and Anti-PT Antibody Concentration Equal to or Above 5 Enzyme-Linked Immunosorbent Assay (ELISA) Units Per Millilitre (EL.U/mL)
Description: Anti-FHA, anti-PRN and anti-PT antibody concentration cut-off value assessed was ≥ 5 ELISA units per millilitre.
Time Frame: Prior to the first dose and one month after the third dose (at study Months 0 and 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 69 | 67 | 71 | 74 | 71
Subjects
  Anti-PT [Month 0] (N=67,62,68,70,69) | 15 | 11 | 18 | 12 | 9
  Anti-PT [Month 3] (N=67,63,69,74,69) | 67 | 63 | 69 | 74 | 69
  Anti-FHA [Month 0] (N=69,63,69,72,70) | 42 | 37 | 42 | 55 | 45
  Anti-FHA [Month 3] (N=67,63,69,74,71) | 67 | 63 | 69 | 74 | 71
  Anti-PRN [Month 0] (N=68,62,71,72,70) | 36 | 25 | 37 | 37 | 37
  Anti-PRN [Month 3] (N=68,67,70,74,71) | 68 | 67 | 70 | 74 | 71

25. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration Equal to or Above 0.15 Microgram Per Millilitre (µg/mL).
Description: Anti-PRP antibody concentration cut-off value assessed was equal to or above (≥) 0.15 microgram per millilitre (µg/mL)
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 41 | 39 | 42 | 42 | 39
Subjects
  Anti-PRP >= 0.15 µg/mL Month 0 (N=41,39,42,42,36) | 39 | 38 | 42 | 42 | 36
  Anti-PRP >= 0.15 µg/mL Month 1 (N=39,39,39,40,39) | 39 | 39 | 39 | 40 | 39

26. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in µg/mL.
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 41 | 39 | 42 | 42 | 39
µg/mL
  Anti-PRP [Month 0] (N=41,39,42,42,36) | 1.306 [0.947 to 1.801] | 1.591 [1.185 to 2.135] | 1.414 [1.068 to 1.871] | 1.764 [1.301 to 2.391] | 0.607 [0.459 to 0.802]
  Anti-PRP [Month 1] (N=39,39,39,40,39) | 36.280 [27.856 to 47.252] | 32.930 [22.797 to 47.567] | 34.107 [24.902 to 46.715] | 47.742 [34.631 to 65.817] | 24.345 [17.445 to 33.974]

27. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titre Equal to or Above 1:128
Description: rSBA-MenC antibody titre cut-off value assessed was ≥1:128
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 42 | 39 | 42 | 41 | 39
Subjects
  rSBA-Menc [Month 0] (N=42,39,41,41,38) | 25 | 24 | 22 | 27 | 26
  rSBA-Menc [Month 1] (N=40,39,42,41,39) | 40 | 36 | 42 | 40 | 39

28. Secondary Outcome: Number of Subjects With Meningococcal Serogroup Y Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenY) Titre Equal to or Above 1:128
Description: rSBA-MenY antibody titre cut-off value assessed was ≥1:128
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 41 | 39 | 42 | 42 | 39
Subjects
  rSBA-MenY [Month 0] (N=41,39,42,42,37) | 24 | 18 | 23 | 6 | 7
  rSBA-MenY [Month 1] (N=40,39,42,40,39) | 40 | 39 | 42 | 6 | 10

29. Secondary Outcome: rSBA-MenC Antibody Titres
Description: Titres are expressed as geometric mean titres (GMTs)
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 42 | 39 | 42 | 41 | 39
Titers
  rSBA-MenC [Month 0] (N=42,39,41,41,38) | 128.0 [74.9 to 218.5] | 144.2 [92.8 to 224.1] | 125.8 [81.0 to 195.3] | 150.6 [96.7 to 234.5] | 195.5 [122.4 to 312.2]
  rSBA-MenC [Month 1] (N=40,39,42,41,39) | 4762.6 [3427.5 to 6617.7] | 2897.7 [1793.1 to 4682.7] | 2626.4 [1893.9 to 3642.3] | 3226.2 [2294.7 to 4535.8] | 11819.3 [8458.6 to 16515.2]

30. Secondary Outcome: rSBA-MenY Antibody Titres
Description: Titres are expressed as geometric mean titres (GMTs)
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 41 | 39 | 42 | 42 | 39
Titres
  rSBA-MenY [Month 0] (N=41,39,42,42,37) | 97.2 [58.4 to 161.8] | 64.0 [37.6 to 108.9] | 100.9 [62.3 to 163.5] | 11.0 [6.3 to 19.1] | 16.1 [8.8 to 29.5]
  rSBA-MenY [Month 1] (N=40,39,42,40,39) | 1708.1 [1313.3 to 2221.4] | 1313.8 [1004.4 to 1718.6] | 1566.0 [1172.8 to 2091.1] | 11.7 [6.8 to 20.2] | 16.5 [8.7 to 31.3]

31. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentration Equal to or Above 0.30 Microgram Per Millilitre (µg/mL)
Description: Anti-PSC antibody concentration cut-off value assessed was ≥0.30 µg/mL
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 38 | 38 | 40 | 40 | 39
Subjects
  Anti-PSC [Month 0] (N=38,38,40,40,38) | 38 | 38 | 40 | 40 | 38
  Anti-PSC [Month 1] (N=33,33,39,37,39) | 33 | 33 | 39 | 37 | 39

32. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentration Equal to or Above 2.0 Microgram Per Millilitre (µg/mL)
Description: Anti-PSC antibody concentration cut-off value assessed was ≥2.0 µg/mL
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 38 | 38 | 40 | 40 | 39
Subjects
  Anti-PSC [Month 0] (N=38,38,40,40,38) | 24 | 30 | 28 | 26 | 27
  Anti-PSC [Month 1] (N=33,33,39,37,39) | 33 | 33 | 39 | 37 | 39

33. Secondary Outcome: Anti-PSC Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in µg/mL.
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 38 | 38 | 40 | 40 | 39
µg/mL
  Anti-PSC [Month 0] (N=38,38,40,40,38) | 2.57 [1.88 to 3.51] | 3.23 [2.55 to 4.08] | 2.53 [2.06 to 3.12] | 3.08 [2.33 to 4.08] | 3.17 [2.46 to 4.08]
  Anti-PSC [Month 1] (N=33,33,39,37,39) | 32.04 [22.99 to 44.65] | 28.00 [19.40 to 40.42] | 19.75 [15.23 to 25.60] | 27.71 [22.23 to 34.54] | 64.41 [50.72 to 81.79]

34. Secondary Outcome: Anti-PSY Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in µg/mL.
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 42 | 39 | 42 | 42 | 38
µg/mL
  Anti-PSY [Month 0] (N=39,39,42,42,38) | 3.72 [2.76 to 5.03] | 5.25 [3.95 to 6.96] | 3.96 [3.02 to 5.19] | 0.16 [0.14 to 0.19] | NA [NA to NA] — Values were below the assay cut-off value of 0.3 µg/mL.
  Anti-PSY [Month 1] (N=42,39,41,40,38) | 26.15 [17.80 to 38.42] | 35.90 [25.33 to 50.88] | 32.18 [25.26 to 40.99] | 0.17 [0.13 to 0.21] | NA [NA to NA] — Values were below the assay cut-off value of 0.3 µg/mL.

35. Secondary Outcome: Number of Subjects With Anti-tetanus Toxoid (Anti-T) Antibody Concentration Equal to or Above 0.1 International Units Per Millilitre (IU/mL).
Description: Anti-tetanus toxoid antibody concentration cut-off value assessed was ≥ 0.1 IU/mL
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 41 | 39 | 42 | 42 | 39
Subjects
  Anti-tetanus [Month 0] (N=41,39,42,42,38) | 41 | 39 | 42 | 42 | 37
  Anti-tetanus [Month 1] (N=39,39,39,40,39) | 39 | 39 | 39 | 40 | 39

36. Secondary Outcome: Anti-T Antibody Concentrations
Description: as for outcome 21
Time Frame: Prior to and one month post booster vaccination (at study Months 0 and 1 - booster phase)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 41 | 39 | 42 | 42 | 39
IU/mL
  Anti-tetanus [Month 0] (N=41,39,42,42,38) | 0.836 [0.655 to 1.067] | 0.986 [0.810 to 1.202] | 0.894 [0.748 to 1.069] | 0.839 [0.693 to 1.016] | 0.322 [0.257 to 0.402]
  Anti-tetanus [Month 1] (N=39,39,39,40,39) | 12.609 [10.769 to 14.762] | 10.175 [8.269 to 12.520] | 9.893 [8.255 to 11.856] | 11.674 [9.538 to 14.288] | 5.474 [4.331 to 6.918]

37. Secondary Outcome: Anti-diphtheria Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in IU/mL.
Time Frame: One month after the third dose (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 68 | 64 | 69 | 74 | 69
IU/mL | 1.016 [0.796 to 1.297] | 0.927 [0.759 to 1.132] | 0.980 [0.788 to 1.219] | 1.012 [0.827 to 1.238] | 1.904 [1.606 to 2.258]

38. Secondary Outcome: Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations
Description: Antibody concentrations are expressed as geometric mean concentrations (GMCs) in milli-International Units per millilitre (mIU/mL).
Time Frame: One month after the third dose (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 62 | 61 | 67 | 72 | 65
mIU/mL | 377.9 [261.7 to 545.8] | 397.0 [271.5 to 580.4] | 408.9 [305.9 to 546.6] | 520.5 [374.1 to 724.3] | 287.3 [194.3 to 424.7]

39. Secondary Outcome: Anti-poliovirus Types 1, 2, 3 Antibody Titres
Description: Titres are expressed as geometric mean titres (GMTs)
Time Frame: One month after the third dose (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 57 | 55 | 58 | 61 | 56
Titers
  Anti-poliovirus type 1 (N=57,55,56,61,56) | 275.5 [206.9 to 366.8] | 242.0 [181.2 to 323.4] | 216.8 [162.6 to 288.9] | 305.2 [229.2 to 406.4] | 282.6 [204.4 to 390.7]
  Anti-poliovirus type 2 (N=55,55,58,61,56) | 155.8 [110.4 to 220.0] | 149.9 [108.3 to 207.7] | 133.7 [95.5 to 187.2] | 123.1 [86.3 to 175.6] | 171.3 [123.2 to 238.1]
  Anti-poliovirus type 3 (N=57,55,58,61,56) | 649.0 [492.3 to 855.7] | 577.2 [418.7 to 795.8] | 451.7 [320.9 to 635.9] | 603.6 [452.7 to 804.6] | 505.7 [375.5 to 681.0]

40. Secondary Outcome: Number of Seroprotected Subjects for Anti-diphtheria Antibodies
Description: Seroprotection status is defined as anti-diphtheria antibody concentrations ≥ 0.1 IU/mL
Time Frame: One month after the third dose (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 68 | 64 | 69 | 74 | 69
Subjects | 66 | 64 | 69 | 74 | 69

41. Secondary Outcome: Number of Seroprotected Subjects for Anti-hepatitis B Antibodies
Description: Seroprotection status is defined as anti-HBs antibody concentrations ≥ 10 mIU/mL
Time Frame: One month after the third dose (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 62 | 61 | 67 | 72 | 65
Subjects | 60 | 60 | 66 | 70 | 61

42. Secondary Outcome: Number of Seroprotected Subjects for Anti-poliovirus Types 1, 2 and 3 Antibodies
Description: Seroprotection status is defined as anti-polio 1, 2 and 3 antibody titres ≥ 1:8
Time Frame: One month after the third dose (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 57 | 55 | 58 | 61 | 56
Subjects
  Anti-poliovirus type 1 (N=57,55,56,61,56) | 57 | 55 | 56 | 61 | 55
  Anti-poliovirus type 2 (N=55,55,58,61,56) | 55 | 55 | 58 | 59 | 56
  Anti-poliovirus type 3 (N=57,55,58,61,56) | 57 | 55 | 58 | 61 | 56

43. Secondary Outcome: Number of Subjects With Vaccine Response to PT, FHA and PRN
Description: Vaccine response rates are defined as appearance of antibodies in subjects who were initially seronegative (i.e., with concentrations < cut-off value) or at least maintenance of pre-vaccination antibody concentrations in subjects who were initially seropositive (i.e., with concentrations ≥ cut-off value), taking into consideration the decreasing maternal antibodies.
Time Frame: One month after the third dose (at study Month 3 - primary phase)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 66 | 62 | 70 | 72 | 70
Subjects
  Anti-PT (N=64,58,66,70,68) | 63 | 58 | 64 | 66 | 68
  Anti-FHA (N=66,59,67,72,70) | 65 | 58 | 65 | 68 | 70
  Anti-PRN (N=66,62,70,72,70) | 61 | 59 | 68 | 63 | 65

44. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling.
Time Frame: During the 8-day (Day 0-7) follow-up period (during the primary phase)
Population: The Total Vaccinated Cohort included all subjects with study vaccine administered for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 78 | 77 | 78 | 78 | 77
Subjects
  Pain | 21 | 20 | 22 | 19 | 19
  Redness | 35 | 38 | 50 | 32 | 46
  Swelling | 31 | 35 | 30 | 27 | 35

45. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Solicited general symptoms assessed were drowsiness, irritability, loss of appetite and fever (fever is defined as rectal temperature ≥ 38.0 degrees Celsius (°C)).
Time Frame: During the 8-day (Day 0-7) follow-up period (during the primary phase)
Population: The Total Vaccinated Cohort included all subjects with study vaccine administered for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 78 | 77 | 78 | 78 | 77
Subjects
  Drowsiness | 39 | 53 | 43 | 37 | 46
  Irritability | 44 | 42 | 51 | 47 | 44
  Loss of appetite | 24 | 34 | 29 | 33 | 30
  Fever (rectal) >= 38.0°C | 25 | 28 | 26 | 28 | 28

46. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Day 0-30) follow-up period (during the primary phase)
Population: The Total Vaccinated Cohort included all subjects with study vaccine administered for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 78 | 77 | 78 | 78 | 77
Subjects | 39 | 33 | 35 | 31 | 26

47. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: Over the full course of the primary phase (up to study Month 3 - primary phase)
Population: The Total Vaccinated Cohort included all subjects with study vaccine administered for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 78 | 77 | 78 | 78 | 77
Subjects | 0 | 1 | 2 | 1 | 3

48. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling.
Time Frame: During the 8-day (Day 0-7) follow-up period (during the booster phase)
Population: The Booster Total Vaccinated Cohort included all subjects who received the booster dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 47 | 42 | 44 | 44 | 44
Subjects
  Pain | 5 | 10 | 8 | 8 | 9
  Redness | 20 | 18 | 22 | 16 | 16
  Swelling | 15 | 12 | 12 | 9 | 10

49. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: as for outcome 45
Time Frame: During the 8-day (Day 0-7) follow-up period (during the booster phase)
Population: The Booster Total Vaccinated Cohort included all subjects who received the booster dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 47 | 42 | 44 | 44 | 44
Subjects
  Drowsiness | 14 | 18 | 18 | 17 | 18
  Irritability | 16 | 18 | 19 | 14 | 17
  Loss of appetite | 11 | 16 | 12 | 10 | 14
  Fever (rectal) >= 38.0°C | 13 | 10 | 16 | 18 | 16

50. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: as for outcome 46
Time Frame: During the 31-day (Day 0-30) follow-up period (during the booster phase)
Population: The Booster Total Vaccinated Cohort included all subjects who received the booster dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 47 | 42 | 44 | 44 | 44
Subjects | 7 | 12 | 13 | 12 | 11

51. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 47
Time Frame: Over the full course of the booster phase (up to study Month 1 - booster phase)
Population: The Booster Total Vaccinated Cohort included all subjects who received the booster dose.
Measure: Number; unit: Subjects
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Number analyzed (Participants) | 47 | 42 | 44 | 44 | 44
Subjects | 1 | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs: Over the full course of the primary and booster phases (up to Month 3 - primary phase and up to Month 1 - booster phase). Unsolicited AEs: During the 31-day (Days 0-30) follow-up period. Solicited AEs: During the 8-day (Days 0-7) follow-up period
Arm/Group | Menhibrix F1/Infanrix-penta Group | Menhibrix F2/Infanrix-penta Group | Menhibrix F3/Infanrix-penta Group | Menitorix/Infanrix-penta Group | Menjugate/Infanrix-hexa Group
Serious Adverse Events (participants affected / at risk) | 1/78 | 1/77 | 2/78 | 1/78 | 3/77
Other Adverse Events (participants affected / at risk) | 70/78 | 71/77 | 73/78 | 71/78 | 70/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Menhibrix F1/Infanrix-penta Group (N=78) | Menhibrix F2/Infanrix-penta Group (N=77) | Menhibrix F3/Infanrix-penta Group (N=78) | Menitorix/Infanrix-penta Group (N=78) | Menjugate/Infanrix-hexa Group (N=77)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Laryngotracheo bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 — Over the full course of the primary phase (up to study Month 3 - primary phase)
Febrile convulsion (Nervous system disorders) | 0/47 | 1/42 | 0/44 | 0/44 | 0/44 — Over the full course of the booster phase (up to study Month 1 - booster phase)
Gastroenteritis (Infections and infestations) | 1/47 | 0/42 | 0/44 | 0/44 | 0/44 — Over the full course of the booster phase (up to study Month 1 - booster phase)
Otitis media (Infections and infestations) | 0/47 | 0/42 | 0/44 | 1/44 | 0/44 — Over the full course of the booster phase (up to study Month 1 - booster phase)
Upper respiratory tract infection (Infections and infestations) | 0/47 | 1/42 | 0/44 | 0/44 | 0/44 — Over the full course of the booster phase (up to study Month 1 - booster phase)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Menhibrix F1/Infanrix-penta Group (N=78) | Menhibrix F2/Infanrix-penta Group (N=77) | Menhibrix F3/Infanrix-penta Group (N=78) | Menitorix/Infanrix-penta Group (N=78) | Menjugate/Infanrix-hexa Group (N=77)
Pain (General disorders) | 21 | 20 | 22 | 19 | 19 — During the 8-day (Day 0-7) follow-up period (during the primary phase)
Redness (General disorders) | 35 | 38 | 50 | 32 | 46 — During the 8-day (Day 0-7) follow-up period (during the primary phase)
Swelling (General disorders) | 31 | 35 | 30 | 27 | 35 — During the 8-day (Day 0-7) follow-up period (during the primary phase)
Drowsiness (General disorders) | 39 | 53 | 43 | 37 | 46 — During the 8-day (Day 0-7) follow-up period (during the primary phase)
Irritability (General disorders) | 44 | 42 | 51 | 47 | 44 — During the 8-day (Day 0-7) follow-up period (during the primary phase)
Loss of appetite (General disorders) | 24 | 34 | 29 | 33 | 30 — During the 8-day (Day 0-7) follow-up period (during the primary phase)
Fever (General disorders) | 25 | 28 | 26 | 28 | 28 — During the 8-day (Day 0-7) follow-up period (during the primary phase)
Upper respiratory tract infection (Infections and infestations) | 11 | 6 | 4 | 8 | 6 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Bronchitis (Infections and infestations) | 6 | 4 | 2 | 3 | 3 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Candidiasis (Infections and infestations) | 6 | 3 | 4 | 2 | 3 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 4 | 4 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1 | 5 | 1 | 4 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 4 | 2 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Pyrexia (General disorders) | 1 | 0 | 4 | 3 | 2 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 4 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 1 | 2 — During the 31-day (Day 0-30) follow-up period (during the primary phase)
Pain (General disorders) | 5/47 | 10/42 | 8/44 | 8/44 | 9/44 — During the 8-day (Day 0-7) follow-up period (during the booster phase)
Redness (General disorders) | 20/47 | 18/42 | 22/44 | 16/44 | 16/44 — During the 8-day (Day 0-7) follow-up period (during the booster phase)
Swelling (General disorders) | 15/47 | 12/42 | 12/44 | 9/44 | 10/44 — During the 8-day (Day 0-7) follow-up period (during the booster phase)
Drowsiness (General disorders) | 14/47 | 18/42 | 18/44 | 17/44 | 18/44 — During the 8-day (Day 0-7) follow-up period (during the booster phase)
Irritability (General disorders) | 16/47 | 18/42 | 19/44 | 14/44 | 17/44 — During the 8-day (Day 0-7) follow-up period (during the booster phase)
Loss of appetite (General disorders) | 11/47 | 16/42 | 12/44 | 10/44 | 14/44 — During the 8-day (Day 0-7) follow-up period (during the booster phase)
Fever (General disorders) | 13/47 | 10/42 | 16/44 | 18/44 | 16/44 — During the 8-day (Day 0-7) follow-up period (during the booster phase)
Upper respiratory tract infection (Infections and infestations) | 5/47 | 6/42 | 4/44 | 2/44 | 4/44 — During the 31-day (Day 0-30) follow-up period (during the booster phase)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.